CLINICAL TRIAL: NCT03601351
Title: Mu Opioid Receptor 1 Expression in Colorectal Cancer and Disease-free Survival Relationship (Morocco). Five-year Follow-up.
Brief Title: MOR-1 Expression in Colorectal Cancer and Disease-free Survival Relationship. Five-year Follow-up.
Acronym: MOROCCO
Status: Completed | Type: Observational
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, PRINCIPAL INVESTIGATOR, Hospital Universitario La Fe
Other Study IDs: ODC-MOR-2018-01
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Cancer
Keywords: CANCER, COLON, OPIOIDS, MOR-1
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TT: Tumor Tissue. Colon or rectum neoplasia stage II and III tumor tissue.
  Interventions: Other: ELISA for MOR-1 expression
- NTT: Nontumorous Tissue. Colon or rectum neoplasia stage II and III adjacent nontumorous tissue.
  Interventions: Other: ELISA for MOR-1 expression

INTERVENTIONS:
Other: ELISA for MOR-1 expression — To evaluate MOR-1 expression differences by immunohistochemical analysis (ELISA - semiquantitative) in paraffin samples from patients with colorectal cancer stage II / III submitted scheduled colorectal surgery between the tumor tissue and the adjacent nontumorous tissue.

SUMMARY:
Colorectal cancer (CRC) is a global burden and one of the most frequent types of cancer. Colorectal cancer therapy is complex and surgery remains the cornerstone for its treatment, combined with chemotherapy and radiotherapy. At diagnosis time, stage II / III is the predominant . There is a growing interest on the potential effect of perioperative anesthetic management on cancer growth and spread. Preclinical studies suggest that opioids could promote direct tumor growth, angiogenesis, metastasis and immunosuppression of cellular and humoral responses, mainly mediated by Mu opioid receptor 1 (MOR-1) activation. Association between increased expression of MOR-1and or perioperative opioids use and shorter DFS or OS has been demonstrated in lung, prostate, gastric and esophagus cancers. Furthermore a pooled analysis suggested that methylnaltrexone, a peripherally acting Mu-opioid receptor antagonist (PAMORA) was associated with increased survival in patients with advanced cancer.

Thus, the expression of the MOR-1 is an indicator of poor prognosis in some cancer types, but its relevance in colon cancer is unknown. The hypothesis of this study is that the increased MOR-1expression in tumor samples from colorectal cancer could be associated to poor disease free survival.

These findings would be of great clinical relevance in order to avoid perioperative opioid use in oncological patients. Moreover PAMORAs could be a valuable tool in perioperative antitumor treatment, since currently these drugs are currently used with confirmed tolerability and low adverse effects in the management of opioid-induced constipation (Opioid Induced Constipation-OIC). Besides MOR 1 expression could constitute a biomarker that guide the investigators to perform neoadjuvant therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To evaluate the association between Mu opioid receptor 1 (MOR-1) expression in patients with colorectal cancer stage II / III submitted to scheduled curative surgery and disease-free survival (DFS) five years follow up after surgery.

SECONDARY OBJECTIVES:

To evaluate the association between the MOR-1 expression in patients with colorectal cancer stage II / III undergoing scheduled curative surgery and overall survival (OS) five years follow up after surgery.

To evaluate the association between MOR-1 expression in patients with colorectal cancer stage II / III submitted to scheduled curative surgery and perioperative complications until postoperative day 28th after surgery.

To evaluate the association between perioperative opioids dose (morphine equivalents) and disease-free survival/overall survival until five years after surgery.

To evaluate MOR-1 expression differences in paraffin samples from patients with colorectal cancer stage II / III submitted scheduled colorectal surgery between the tumor tissue and the adjacent nontumorous tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Colorectal scheduled surgery between January 2010- December 2013.
* Colon / rectum neoplasia Stage II / III (T3 / T4 N + M0).

Exclusion Criteria:

* Stage I or Stage IV
* Non-oncological colorectal surgery
* Non-elective surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled colorectal surgery stage II / III for primary colorectal cancer between 01/01/2010 from 31/12/2013.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Expression of MOR1. | Six months
  Immunohistochemical analysis (ELISA - semiquantitative) to asses expression of MOR1 in tumor tissue and adjacent nontumorous tissue.
Disease free survival. | Five years.
  Disease free survival 5 years after surgery.

SECONDARY OUTCOMES:
Local recurrence. | Five years.
  Five years follow up after surgery.
Lymphatic relapse. | Five years.
  Five years follow up after surgery.
Metastasis. | Five years.
  Reproduction or extension of the tumor to another part of the body. Five years follow up after surgery.
Type of recurrence (local, regional or distant). | Five years.
  Five years follow up after surgery.
Overall Survival. | Five years.
  Five years follow up after surgery.
Morphine equivalents. | During surgery and up to 96 hours during the perioperative period.
  Morphine equivalents consumption during perioperative period.
Perioperative complications. | 28 days.
  Perioperative complications until postoperative day 28th.

CONTACTS AND LOCATIONS:
Overall Officials: OSCAR DIAZ-CAMBRONERO, MD, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Hospital Universitario La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided